CLINICAL TRIAL: NCT02524639
Title: Pilot Study of the Efficacy and Safety of Sirolimus in the Treatment of Congenital Hyperinsulinism.
Brief Title: Sirolimus for the Treatment of Hyperinsulinism
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to strict inclusion and exclusion criteria no subjects were enrolled
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Diva De Leon, Study Principal Investigator, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-011973
Record Dates: First submitted 2015-08-12; First posted 2015-08-17 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Hyperinsulinism
MeSH Terms: conditions — Hyperinsulinism | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus (Experimental): All enrolled subjects will receive Sirolimus 1 mg/m2/day twice a day for 6 weeks.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Subjects will receive 1 mg/m2/day orally for 6 weeks. Maintenance dose will be titrated up or down by 0.25-0.5 mg/m2/day every 4 days. Serum concentration will be checked on day 4 after initial therapy and 4 days after any dose adjustment. Levels will be checked at lease once a week during the duration of the study. Target serum concentration range is 5-10 ng/mL.
  Other Names: Rapamune

SUMMARY:
The purpose of this pilot study is to generate data to assess feasibility of study design/procedures and for formal sample size estimation for a larger multicenter study of the efficacy and safety of sirolimus in infants with medically-unresponsive congenital hyperinsulinism (HI) due to inactivating mutations of adenosine triphosphate-sensitive potassium (KATP) channels.

DETAILED DESCRIPTION:
Treatment options for children with diffuse adenosine triphosphate-sensitive potassium (KATP) channel hyperinsulinism (KATPHI) are limited and most of them require a near-total pancreatectomy to control the hypoglycemia. However, at least 40% of these children continue to have persistent hypoglycemia after surgery and their long-term outcomes are complicated by the development of diabetes.

There is evidence that suggests that mammalian target of rapamycin (mTOR) inhibitors are useful in controlling the hypoglycemia in hyperinsulinemic hypoglycemia. But before adapting this as standard therapy for children with hyperinsulinism, a carefully controlled study of the efficacy and safety of sirolimus for hyperinsulinism is clearly needed.

Sirolimus is an mTOR inhibitor, which is FDA-approved for the prophylaxis of organ rejection in patients age 13 years and older receiving kidney transplantation. This is an open label pilot study to assess the effect, safety and tolerability of sirolimus in infants with diazoxide-unresponsive HI due to mutations in the genes encoding the KATP channels. Subjects will be treated with sirolimus for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age ≥14 days to 12 months.
2. Confirmed diagnosis of hyperinsulinism.
3. Mutation analysis results demonstrating bi-allelic mutations in either ABCC8 or KCNJ11.
4. Failure to respond to maximal dose of diazoxide (15 mg/kg/day), if diazoxide is indicated.

   1. Unable to wean intravenous dextrose after at least 3 days of diazoxide therapy and/or
   2. Persistent hypoglycemia after at least 3 days of diazoxide therapy
5. High glucose infusion rate requirement (greater or equal to 10 mg/kg/min).
6. Parental/guardian permission (informed consent).

Exclusion Criteria:

1. Infants with suspected or confirmed focal hyperinsulinism who are candidates for surgical resection
2. Current therapy with diazoxide. Subjects may be eligible for participation 48 hrs after discontinuation of diazoxide.
3. Laboratory abnormalities that indicate clinically significant hematologic, hepatobiliary, or renal disease:

   1. AST/SGOT > 2.5 times the upper limit of normal
   2. ALT/SGPT > 2.5 times the upper limit of normal
   3. Total bilirubin > 2.5 times the upper limit of normal
   4. Hemoglobin < 9 gm/dL
   5. White blood cell count < 3,000/ mm3
   6. Platelet count < 100,000/mm3
   7. Creatinine > 2.5 times the upper limit of normal
4. Evidence of active infection.
5. Evidence of cardiac or respiratory failure.
6. Known immune deficiency.
7. Preterm (< 37 week gestation at birth).
8. Treatment with immunosuppressants.
9. Treatment with any drug known to interact significantly with sirolimus (strong inducers and strong inhibitors of CYP3A4 and P-gp with risk category D and X) including:

   Cyclosporine, clozapine, conivaptan, crizotinib, dabrafenib, dipyrone, boceprevir, echinacea, efavirenz, enzalutamide, fluconazole, fosphenytoin, fusidic acid, idelalisib, leflunomide, lomitapide, mifepristone, mitotane, natalizumab, nelfinavir, phenytoin, pimecrolimus, pimozide, posaconazole, roflumilast, St Johns Wort, stiripentol, tacrolimus, telaprevir, tofacitinib, rifampin, rifabutin, ketoconazole, voriconazole, itraconazole, erythromycin, telithromycin, clarithromycin
10. Any investigational drug use within 5 half-lives of the drug prior to initiation of therapy.

    Subjects who had participated in other investigational drug studies will be eligible to participate after 5 half-lives from the last dose of the investigational agent and have recovered from acute investigational agent associated toxicity
11. History of surgical procedure within 8 weeks of enrollment.
12. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-08-12 (Estimated); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Number of children off intravenous dextrose support | 6 weeks

SECONDARY OUTCOMES:
Change in number hypoglycemic episodes per child per day | 6 weeks
Plasma insulin levels during fasting | 8 hours
Number of participants with Adverse Events | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diva De Leon, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States